CLINICAL TRIAL: NCT00000663
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant CD4 Immunoglobulin G (rCD4-IgG) in Infants and Children With Documented HIV-1 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ACTG 139; D0172g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Injections, Intravenous; IgG; Drug Evaluation; Acquired Immunodeficiency Syndrome; Antigens, CD4; Carrier Proteins
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — CD4 Immunoadhesins

INTERVENTIONS:
Drug: CD4-IgG

SUMMARY:
To determine the safety profile, assess pharmacokinetic properties (blood levels), and obtain preliminary indication of the antiviral and immunologic effects of recombinant CD4 immunoglobulin G (CD4-IgG).

CD4-IgG may be effective in blocking HIV transmission and spread, that is, CD4-IgG has antiviral effects. Studies done in adult patients with AIDS and AIDS related complex (ARC) have shown that rCD4 can be safely administered by intravenous bolus, intramuscular or subcutaneous injection. No serious or dose-limiting, drug-related toxicities have been observed to date.

DETAILED DESCRIPTION:
CD4-IgG may be effective in blocking HIV transmission and spread, that is, CD4-IgG has antiviral effects. Studies done in adult patients with AIDS and AIDS related complex (ARC) have shown that rCD4 can be safely administered by intravenous bolus, intramuscular or subcutaneous injection. No serious or dose-limiting, drug-related toxicities have been observed to date.

Patients receive one intravenous injection the first week, followed by a 6 day washout period and then intravenous injections on a twice weekly basis from week 2 to week 12. The dose per injection may vary. The study evaluates 2 groups: (1) Children 3 months to 5 years of age; (2) Infants 0-3 months of age.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* HIV-1 infection, or if less than 15 months old, born to mother with HIV-1 infection.
* Legally qualified guardian with the ability to sign a written, informed consent form.
* Willingness to abstain from all other experimental therapy for HIV-1 infection during the first 12 weeks of the study period.
* Anticipated life expectancy of at least 3 months.

Prior Medication:

Allowed:

* Prophylactic anti-Pneumocystis carinii pneumonia (PCP) or antifungal therapy.
* Gamma globulin as prophylaxis for measles and varicella.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Past or present history of neurological abnormalities including withdrawal syndrome or seizures.
* Past or present history of any serious active opportunistic infection including Pneumocystis carinii pneumonia (PCP).
* Echocardiogram values > 2 standard deviations from normal.
* Hematologic, renal, or hepatic insufficiency.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Intravenous gamma globulin (IVIG) except as prophylaxis for measles and varicella.
* Cancer chemotherapy.
* Corticosteroids.
* Other known immunomodulatory agents.
* Other experimental therapy not specifically allowed.

Patients with the following are excluded:

* Hematologic, renal, or hepatic insufficiency.
* Past or present history of any serious active opportunistic infection.

Prior Medication:

Excluded for a minimum of 3 weeks prior to study entry:

* Zidovudine (AZT).
* Intravenous gamma globulin (IVIG).
* Cancer chemotherapy.
* Immunomodulatory agents.
* Acyclovir and other experimental therapy.

Risk Behavior:

Excluded:

* Patients born to substance abusing mothers (including alcohol) during the pregnancy.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18

CONTACTS AND LOCATIONS:
Overall Officials: R Yogev, Study Chair; W Shearer, Study Chair
Locations (7):
- United States (7):
  - UCSD Treatment Ctr, San Diego, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Cook County Hosp, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - North Shore Univ Hosp, Great Neck, New York
  - Columbia Univ Babies' Hosp, New York, New York
  - Texas Children's Hosp / Baylor Univ, Houston, Texas

REFERENCES:
- [Background] Weintrub P, Yogev R, Conner E, Wilfert K, Mordenti J, Ammann AJ. Safety and pharmacokinetics of recombinant CD4 in children with HIV infection. Int Conf AIDS. 1990 Jun 20-23;6(2):95 (abstract no FB23)
- [Background] Shearer WT, Israel RJ, Starr S, Fletcher CV, Wara D, Rathore M, Church J, DeVille J, Fenton T, Graham B, Samson P, Staprans S, McNamara J, Moye J, Maddon PJ, Olson WC. Recombinant CD4-IgG2 in human immunodeficiency virus type 1-infected children: phase 1/2 study. The Pediatric AIDS Clinical Trials Group Protocol 351 Study Team. J Infect Dis. 2000 Dec;182(6):1774-9. doi: 10.1086/317622. Epub 2000 Oct 27. PMID 11069253